CLINICAL TRIAL: NCT05698355
Title: Telerehabilitation in Chronic Pelvic Pain
Acronym: CPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Alime Buyuk, Principal Investigator, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Akdeniz
Record Dates: First submitted 2023-01-16; First posted 2023-01-26 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Pelvic Pain; Telerehabilitation; Pelvic Floor; Relaxation
MeSH Terms: conditions — Pelvic Pain

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation group (Experimental): Multimodal self-treatment-based telerehabilitation will be implemented with a video conference method. For telerehabilitation, at each session, manual therapy techniques, (i.e., stretching, myofascial release, and tissue desensitization), sex education, and pelvic floor muscle relaxation massages with a pelvic wand (i.e., relaxation, stretching) using small intra-vaginal wand were used. Women were also asked to perform home exercises resembling those performed under supervision five times per week as well as auto-insertion exercises with a pelvic wand in addition to desensitization techniques three times per week.
  Sessions consist of 60 minutes. Telerehabilitation will take place 2 days a week for 12 weeks.
  Interventions: Other: Telerehabilitation Treatment
- Education group (No Intervention): 60 minutes of video recording training will be given about pelvic pain relaxation exercises.

INTERVENTIONS:
Other: Telerehabilitation Treatment — Telerehabilitation includes self-massages for pelvic floor muscle, sex education, breathing, myofascial releasing with wand, and pelvic floor relaxing exercises.
  Arms: Telerehabilitation group

SUMMARY:
Objective: Physical therapists utilize telerehabilitation as the common term for telehealth applications. Many physiotherapists worked as telehealth providers during the coronavirus pandemic. The objective of the study will show the efficacy of Telerehabilitation-Based Physical Therapy (TBPT) on pain intensity and treatment satisfaction in patients with chronic pelvic pain.

Method: This study is a prospective study of patients with chronic pelvic pain.42 participants will include the study. Patients who have any other distribution pattern of pelvic pain were equally considered for therapy. Women age between 18-50 years will be include. Their symptoms should be one of these follows such as chronic pain in pelvic region, hyperalgesia in vulva, and pain during sitting or intercourse. They will get diagnosed by a gynecologist who is a multidisciplinary team comprising and referred to a pelvic health physiotherapist. Prior to treatment patients will complete questionnaires and interview a pelvic health physiotherapist. Pain symptoms will be assessed with the Visual Analog Scale (VAS) and The Pelvic Pain Impact Questionnaire (PPIQ) before and after treatment. Patient Global Impression of Improvement (PGI-I) for evaluating patient satisfaction after treatment. Women with chronic pelvic pain will be treated for 16 sessions (an hour for each session) in 8 weeks with the TBPT technique by the same pelvic health physiotherapist (AB). Patients will apply internal and external trigger point release therapy and self-massage techniques by themselves with Telerehabilitation-Based Physical Therapy.

DETAILED DESCRIPTION:
Telerehabilitation is described as the remote conveyance of healthcare services and clinical information using information and telecommunication technologies involving the internet, wireless satellite, and telephone media to provide a series of rehabilitation services by eliminating the barriers of distance, time, and travel to receive care. There is an abundance of commercially available applications (such as Zoom) offered for health care monitoring and management. Most of the studies have employed telerehabilitation methods with patients who have pain, mainly for assessment or exercise programs. There is not any study on the telerehabilitation application of physical therapy in patients with chronic pelvic pain during the coronavirus pandemic.

Our conceptual framework is based on two arguments. First, physiotherapists need physical access to their patients only for a limited number of interventions. Most of the methods used by physiotherapists to treat their patients can be conducted at a distance without having direct access to the patient. Previous studies have shown that telerehabilitation can be used in many cases and provide results on par with face-to-face treatment. In fact, self-administered treatment was found to be effective even in the case of postal treatment where the participants received instruction through postal systems.

Second, the pelvic floor area is relatively well-suited for self-treatment. Most, if not all, of the exercises and procedures, can be safely conducted by the patients themselves. The patients can even use pelvic wands and dilators for harder-to-reach inner release points. Therefore, training the patient and supervising and guiding self-administered procedures should be sufficiently effective to reduce pelvic pain and reach patient satisfaction in most cases.

The aim of the study will show the efficacy of Telerehabilitation-Based Physical Therapy (TBPT) on pain intensity and treatment satisfaction in patients with chronic pelvic pain.

ELIGIBILITY:
Inclusion Criteria:

* experienced pelvic pain (dyspareunia) for over six (6) months prior to the study
* to be able to use the internet and their willingness to participate.
* no pelvic floor surgeries
* no C-section and birth history
* to have a diagnoses by dyspareunia

Exclusion Criteria:

* to have endometriosis
* to have a pelvic health physiotherapy history
* pelvic organ prolapse, or a previous pelvic organ surgery.
* the use of analgesics in the previous three (3) months,
* to have a pregnancy,
* to have an active vaginal or urinary tract infection, or suffering from other comorbidities that affect the lower urinary tract such as diabetes mellitus

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Pelvic Pain Impact Questionnaire | 1-3 monts
  The Pelvic Pain Impact Questionnaire is a questionnaire composed of eight (8) questions. The patient is asked to grade how pelvic pain has affected various activities on a 5-point Likert scale. The total score is obtained by adding the scores given for each item, a high score is directly proportional to the severity of pain.
VAS | 1-3 months
  The VAS is frequently used in cases where rapid measurement of pain intensity is required in clinical and laboratory conditions. It consists of drawing a line from zero (0) to ten (10) and ask the patient to mark the pain intensity on the line where zero (0) means "I have no pain" and ten (10) means "the most severe pain possible".
The Female Sexual Function Index | 1-3 months
  The Female Sexual Function Index is a brief multidimensional scale for assessing sexual function in women. The scale has received initial psychometric evaluation, including studies of reliability, convergent validity, and discriminant validity
The Female Sexual Distress Scale-Revised | 1-3 months
  The Female Sexual Distress Scale-Revised was used to assess sexual distress, with higher scores relating to more sexual distress
Vaginal Penetration Cognition Questionnaire | 1-3 months
  To assess cognition regarding vaginal penetration in women with vaginismus or dyspareunia

SECONDARY OUTCOMES:
The Patient Global Impression of Change | 1-3 motnhs
  The Patient Global Impression of Change allowed the participants to self-report their perceived improvement (categories ranging from very much improved to very much worse). The PGI-I requires the patient to grade on a seven (7) point likert scale how the condition has evolved compared to how it was prior to the treatment. All questionnaires have validity and reliability in Turkish language .

CONTACTS AND LOCATIONS:
Overall Officials: Alime Buyuk, Principal Investigator — Akdeniz University
Locations (1):
- Alime Buyuk, Antalya, Select State / Province...a, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Padoa A, McLean L, Morin M, Vandyken C. The Overactive Pelvic Floor (OPF) and Sexual Dysfunction. Part 2: Evaluation and Treatment of Sexual Dysfunction in OPF Patients. Sex Med Rev. 2021 Jan;9(1):76-92. doi: 10.1016/j.sxmr.2020.04.002. Epub 2020 Jul 4. PMID 32631813
- [Background] Morin M, Dumoulin C, Bergeron S, Mayrand MH, Khalife S, Waddell G, Dubois MF; PVD Study Group. Multimodal physical therapy versus topical lidocaine for provoked vestibulodynia: a multicenter, randomized trial. Am J Obstet Gynecol. 2021 Feb;224(2):189.e1-189.e12. doi: 10.1016/j.ajog.2020.08.038. Epub 2020 Aug 18. PMID 32818475
- [Background] Cyr MP, Dostie R, Camden C, Dumoulin C, Bessette P, Pina A, Gotlieb WH, Lapointe-Milot K, Mayrand MH, Morin M. Improvements following multimodal pelvic floor physical therapy in gynecological cancer survivors suffering from pain during sexual intercourse: Results from a one-year follow-up mixed-method study. PLoS One. 2022 Jan 25;17(1):e0262844. doi: 10.1371/journal.pone.0262844. eCollection 2022. PMID 35077479
- [Background] Cyr MP, Dumoulin C, Bessette P, Pina A, Gotlieb WH, Lapointe-Milot K, Mayrand MH, Morin M. Feasibility, acceptability and effects of multimodal pelvic floor physical therapy for gynecological cancer survivors suffering from painful sexual intercourse: A multicenter prospective interventional study. Gynecol Oncol. 2020 Dec;159(3):778-784. doi: 10.1016/j.ygyno.2020.09.001. Epub 2020 Oct 1. PMID 33010968